CLINICAL TRIAL: NCT02953522
Title: Polymorphism C677T MTHFR and Diet With Folate in Oxidative Stress, Lipid Profile and Homocysteine
Brief Title: Polymorphism C677T MTHFR and Effects of Folate Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Marina Ramalho Ribeiro, Nutritionist and Master Degree Student of Science of Nutrition, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUParaíbaa
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Overweight and Obesity
Keywords: Polymorphism; Folate; Oxidative stress; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 191 mcg/day of Folate (Other): Diet with 191 mcg/day of Folate
  Interventions: Other: 191 mcg/day of Folate
- 90 mcg/day of Folate (Other): Diet with 90 mcg/day of Folate
  Interventions: Other: 90 mcg / day of Folate

INTERVENTIONS:
Other: 191 mcg/day of Folate — Diet containing 191 mcg / day of Folate
  Arms: 191 mcg/day of Folate
Other: 90 mcg / day of Folate — Diet containing 90 mcg / day of Folate
  Arms: 90 mcg/day of Folate

SUMMARY:
The C677T polymorphism in the MTHFR gene is related to several significant biochemical changes, as dyslipidemia, changes in serum levels of homocysteine, folic acid, vitamin B12 and some oxidative stress markers such as the CAT and MDA, leading to a high risk of the emergence of cardiovascular disease (CVD). A diet containing antioxidants, especially folate, is characterized by being beneficial for individuals with this genetic alteration to possess anti-inflammatory function, act on and oxidative stress play an important gene function. The aim of this study was to evaluate the influence of the C677T polymorphism of the MTHFR gene and the effect of a diet containing folate on oxidative stress, lipid profile and homocysteine levels in adult women are overweight or obese. This is an intervention study, double-blind, held in a city in northeastern Brazil. The study included 48 adult women (20-59 years old) with BMI of 26.19 kg / m² and 49.64 kg / m², in which we evaluated the CAT levels, MDA, lipid profile, folic acid, homocysteine and vitamin B12 addition genotyping for the C677T polymorphism in the MTHFR gene and the food consumption by the food recall 24 hours, being divided by randomization into two groups received daily for 8 weeks, 300g vegetables rich in folate containing 191 ug and 90 ug of this nutrient.

DETAILED DESCRIPTION:
This work is linked to a population-based survey entitled "Diagnosis and Intervention II Cycle Situation Food, Nutrition and Noncommunicable Diseases prevalent over the city of João Pessoa Population / PB" (II DISANDNT / PB). For the realization of this dissertation home visits and the questionnaires related to anthropometric and food intake assessment were conducted by teams of undergraduate researchers and graduates of Nutrition Course, masters and doctoral students of the Post Graduate Program in Nutrition Sciences (PPGCN) of UFPB duly previously trained at the beginning of data collection and after completion of the pilot study.

After the selection of individuals from the sample of adults who participated in the II DISANDNT / JP and considering the inclusion criteria and genotyping of the C677T polymorphism in the MTHFR gene, they were invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adult women, aged 20 to 59, sound overweight or obese
* Individuals of different socioeconomic conditions
* Users or not drugs
* Cognitive state preserved and accept participate

Exclusion Criteria:

* Drinkers, smokers or neuropsychiatric disorders
* Users drugs known to interfere with the metabolism of folic acid (the last 3 months), as prednisone, hydrocortisone, dexamethasone, chloramphenicol, acetylsalicylic acid
* Multivitamin supplement users, minerals, appetite suppressants and steroids
* Individuals with chronic diseases with influence on the endocrine and metabolic system
* Pregnant or planning to become pregnant during the study period

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in value of total antioxidant capacity | 8 weeks
  Change in value of total antioxidant capacity

CONTACTS AND LOCATIONS:
Overall Officials: Maria José Carvalho Costa, Doctor, Study Director — UFPB

IPD SHARING:
Plan to Share IPD: Yes
The data of the participants are in the excel database